CLINICAL TRIAL: NCT03207945
Title: Effect of PCSK9 Inhibition on Cardiovascular Risk in Treated HIV Infection (EPIC-HIV Study)
Acronym: EPIC-HIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Priscilla Hsue, MD, Professor of Medicine, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-22800
Record Dates: First submitted 2017-06-28; First posted 2017-07-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Dyslipidemias; Cardiovascular Diseases; HIV Infections
MeSH Terms: conditions — Dyslipidemias; Cardiovascular Diseases; HIV Infections | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alirocumab (Experimental): Patients randomized into the alirocumab arm will start off with 75 mg alirocumab administered every two weeks for two doses and will be upwardly titrated to 150 mg alirocumab if subjects demonstrate LDL ≥ 50 mg/dL at week 4. Subjects demonstrating LDL-C <50mg/dl will remain on the same 75mg dose throughout the trial.
  Interventions: Drug: Alirocumab
- Placebo (Placebo Comparator): Patients randomized into the placebo arm will receive 75 mg or 150 mg or placebo administered once every two weeks throughout the trial
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alirocumab — Alirocumab (Sar236553/REG 727) is a fully humanized monoclonal antibody against the proprotein convertase subtilisin kexin type 9 (PCSK9) enzyme responsible for the degradation of the low-density lipoprotein receptor (LDLR), and is developed by Regeneron Pharmaceuticals/Sanofi.
  Other Names: Sar236553/REG727
  Arms: Alirocumab
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Atherosclerosis in the setting of HIV infection is distinct and includes increased vascular inflammation, worsened endothelial function, and a predominance of non-calcified plaque. These outcomes can be assessed using specialized noninvasive imaging which strongly predict future CV events in the general population.

PCSK9 has emerged as an important pharmacologic target for cholesterol lowering in the general population and recent studies among individuals without HIV have shown that PCSK9 inhibitor therapy is safely tolerated and significantly reduces major CV events in the general population.

The investigators will perform a clinical trial of PCSK9 inhibition in the setting of HIV infection. This will be a randomized, placebo-controlled study to evaluate the effects of PCSK9 inhibition on vascular inflammation, endothelial function, and non-calcified plaque using a PCSK9 inhibitor called alirocumab. This study will recruit 140 treated individuals with HIV who are aged 40 and older, with known CVD or risk factors for CVD and who have evidence of vascular inflammation at baseline.

The primary and secondary objective of this study is to determine whether PCSK9 inhibition can improve arterial inflammation as assessed by FDG-PET/CT and endothelial function as assessed by flow mediated vasodilation. The investigators will correlate changes in arterial inflammation and endothelial function with lipids and markers of inflammation and immune activation.

The tertiary objective is to perform a pilot evaluation of the impact of PCSK9 inhibition on non-calcified plaque as measured by coronary CT angiography. Non-calcified plaque measurements will be correlated with changes in lipid parameters and markers of inflammation and immune activation.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) due to atherosclerosis continues to be the leading single cause of death in industrialized countries. High serum lipid levels, and especially high low-density lipoprotein cholesterol (LDL-C) levels, have been demonstrated to strongly and directly correlate with CVD risks by numerous epidemiological studies. Moreover, large prospective clinical outcome trials have demonstrated that lowering LDL-C decreases cardiovascular morbidity and mortality. A meta-analysis of 26 randomized clinical trials comprising 170,000 participants showed that more intensive statin therapy compared to less intensive regimens will reduce coronary deaths or myocardial infarction by an additional 13%.

HIV-infected individuals represent a unique and increasing subset of atherosclerosis. With the advent of antiretroviral therapy, HIV-infected individuals now have much improved survival and are faced with health issues related to aging, including cardiovascular disease. Individuals with HIV have higher rates of coronary events compared to controls even in the setting of treated and suppressed disease and a growing body of literature suggests that they are at increased risk for myocardial infarction, atherosclerosis, and sudden cardiac death. Many facets of atherosclerosis differ in HIV-infected individuals compared to uninfected individuals with atherosclerosis. HIV-infected patients with acute coronary syndromes are younger and more likely to be males and smokers, with low high density lipoprotein-cholesterol (HDL-C), compared to other acute coronary syndrome patients. With respect to pathophysiology, viral replication, antiretroviral drugs all contribute to atherosclerosis.

HIV-associated inflammation induces pro-atherogenic lipid abnormalities and anti-retroviral therapy leads to the development of metabolic abnormalities such as dyslipidemia, lipodystrophy and insulin resistance. In a large cross-sectional study, 27% of subjects receiving combination therapy including a protease inhibitor had a total cholesterol level exceeding 240 mg/dl, compared to 8% of untreated HIV subjects, and 40% had triglyceride levels above 200 mg/dl, compared to 15% in untreated subjects. The prevalence and severity of dyslipidemia varies among different antiretroviral drugs; however, hypertriglyceridemia and low HDL-cholesterol were associated with HIV infection even before the advent of antiretroviral therapy. Total, HDL-C, and LDL-C decrease at the time of HIV infection, and with antiretroviral treatment total and LDL-C levels increase to pre-infection levels while HDL-C remains low.

Abnormalities in body composition have been reported in 40-50% of HIV-infected patients, with higher rates in those receiving combination antiretroviral therapies. Subcutaneous lipoatrophy commonly affects the face, limbs, and buttocks, and is accompanied by central fat accumulation. Hyperinsulinemia is often also present. In a representative study, diabetes was present in 7% of HIV-infected adults with fat accumulation or lipoatrophy, as compared to 0.5% of control subjects matched for age and BMI. The corresponding rates of glucose intolerance were 35% and 5% respectively. Compared to healthy control subjects, HIV-infected men treated with combination antiretroviral therapy were 4 times as likely to develop diabetes over a 3-year observation period.

The increased cardiovascular risk and dyslipidemia in HIV-infected individuals is difficult to treat for several reasons. Statins reduce LDL-C levels less in HIV-infected individuals compared to uninfected controls. Fibrates reduce triglyceride levels less in HIV-infected individuals compared to uninfected controls as well. Drug-drug interactions between statins and protease inhibitors increase the risk of adverse events. Due to these interactions, simvastatin and lovastatin are contraindicated among individuals receiving protease inhibitors and the dose of atorvastatin should not exceed 40 mg. Even interactions with rosuvastatin, which is not metabolized by the cytochrome P450 system, have been described.

As a consequence, physicians may avoid treating HIV-infected individuals who would benefit from statins, or use lower doses or less potent statins, reducing the potential for cardiovascular event reduction. High triglyceride levels in HIV-infected subjects are common, and the combination of a fibrate plus antiretroviral therapy increases the risk of drug-drug adverse events, even before consideration of a statin.

Statin treatment reduces lipid levels modestly in HIV subjects. Among 72 HIV-infected subjects in the SATURN-HIV trial randomized to rosuvastatin 10 mg/day, LDL-C was reduced by 25.3% by week 24. In another study, of 83 HIV-infected subjects, rosuvastatin 10 mg and pravastatin 40 mg/day reduced LDL-C by 37% and 19% respectively at 45 days. Among 151 HIV-infected subjects randomized to rosuvastatin 10 mg, atorvastatin 10 mg, or pravastatin 40 mg/day, LDL-C reductions were greater with rosuvastatin at this dose, but all 3 statins significantly and similarly reduced serum levels of hs-CRP and TNF-a.

Approximately 1/3 of individuals with HIV-infection are co-infected with hepatitis C. Elevated hepatic enzymes due to hepatitis C represent a relative contraindication to statin therapy, and some evidence suggests that a statin might increase hepatitis C activity. Finally, HIV-infected patients often need many medications and have a large daily pill burden. Compliance suffers, but has been shown to improve when single tablet regimens reduce daily pill load. Long-acting injectable antiretroviral drugs are under development as a strategy to reduce pill burden and improve compliance. PCSK9 inhibitor injections would dovetail well with this approach. For these reasons, PCSK9 inhibitor therapy offers advantages over statin therapy in this unique population.

That statins might favorably influence the evolution of atherosclerosis in HIV-infected subjects is suggested by a recent trial where 40 HIV subjects with mild coronary atherosclerosis by CT angiography and aortic inflammation by FDG-PET imaging were randomized to atorvastatin 20-40 mg/day or placebo and were followed for 12 months. Atorvastatin significantly reduced non-calcified coronary plaque volume relative to placebo, as well as the number of high-risk plaques.

In the HIV-uninfected population, statin therapy produced significant and rapid dose-dependent reductions in FDG update that were reflective of changes in atherosclerotic plaque inflammation. In addition, lipoprotein apheresis resulted in significant reduction of arterial inflammation. Recently, addition of evolocumab was found to result in a greater decrease in percent atheroma volume using intravascular ultrasound. All of these studies which were performed in the non-HIV population provide a strong scientific rationale for studying the role of PCSK9 inhibition in HIV. Namely, given the strong association between HIV, noncalcified plaque, and arterial inflammation, PCSK9 therapy may play a unique role in reducing HIV-associated atherosclerosis, Alirocumab (Sar236553/REG 727) is a fully humanized monoclonal antibody against the proprotein convertase subtilisin kexin type 9 (PCSK9) enzyme responsible for the degradation of the low-density lipoprotein receptor (LDLR), and is developed by Regeneron Pharmaceuticals/Sanofi. In a randomized trial of 2341 patients with heterozygous familiar hypercholesterolemia or with established coronary heart disease or a CHD risk equivalent with LDL levels≥70mg/dL and were receiving treatment with statins at the maximum tolerated dose with or without other lipid-lowering therapy. Patients were randomly assigned to a 2:1 ratio to receive alirocumab 150mg or placebo every 2 weeks for 78 weeks. At week 24 the difference between the alirocumab and placebo groups from baseline to calculated LDL was -62 percentage points. The alirocumab group had higher rates of injection site reactions, myalgia, neurocognitive events and ophthalmologic events. The rate of major adverse cardiovascular events was lower in the alirocumab group as compared to placebo in a post hoc analysis (p=0.02).

Preliminary data on 6 HIV-infected individuals inadvertently enrolled in a PCSK9 inhibitor study using evolocumab demonstrated that LDL was lowered 60%, along with significant reductions in triglycerides and Lp(a) and was well tolerated (unpublished data)

Based on these findings a dose of 75 mg every 2 weeks for 6 weeks followed by an upward titration to 150 mg every 2 weeks for those with LDL-C >50 mg/dl for the remainder of the study for this trial will be used. Based on population PK/PD modeling, a dose of 150 mg every 2 weeks in patients on a background of statins is estimated to be equivalent to approximately 80% of the maximal response for LDL-C lowering (-67%). Assuming an average LDL C at baseline of 100 mg/dL for HIV-infected individuals, the mean absolute LDL-C reduction is predicted to be approximately -60 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
2. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Males and females equal or greater than 40 years of age.
4. Documented HIV infection.
5. HIV-1 RNA level below 200 copies/mL for at least 12 weeks prior to study entry
6. CD4 T Cells ≥200 cells/mm3 at screening
7. Continuous ART for at least 12 weeks with no change in regimen prior to study entry.
8. Moderate or high CVD risk defined as: documented CVD as assessed by meeting at least 1 of 3 criteria below:

   1. Coronary artery disease (CAD)
   2. Cerebrovascular disease
   3. Peripheral arterial disease

   OR any one of the following CVD risk factors:
   1. Controlled type II diabetes mellitus (HbA1C ≤ 8.0%)
   2. Family history: a first degree relative who had a heart attack, stroke, or documented CVD as defined in the previous section that occurred: a. When they were age 55 years or younger for males (father, uncle, or brother) b. When they were age 60 years or younger for females (mother, aunt, or sister)
   3. Current smoking
   4. Hypertension
   5. Dyslipidemia
   6. A hsCRP ≥ 2mg/L at screening.
9. Lipids at screening visit:

   * Fasting LDL-C ≥ 70 mg/dL (1.81 mmol/L);
   * Fasting TG ≤ 600 mg/dL (6.78 mmol/L).
10. If subjects meet ACC/AHA criteria for statin therapy and are not currently on a statin, subjects must be taking a stable dose of statin for at least 4 weeks, unless they are statin intolerant, refuse to take a statin, or have a medical condition (e.g. chronic hepatitis) where a statin is contraindicated.

Exclusion Criteria:

1. Subjects who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Regeneron employees.
2. Participation in other studies involving small molecule investigational drug(s).
3. Subjects who are unable to receive injections, as either a self-injection, or administered by another person.
4. Subjects requiring daily insulin therapy
5. Intended modification of ART in the next 52 weeks
6. History of a cardiovascular or cerebrovascular event or procedure (e.g., myocardial infarction, stroke, transient ischemic attack, angioplasty) during the past 90 days.
7. Congestive heart failure, New York Heart Association functional class IV, or left ventricular ejection fraction measured by imaging known to be <25%. (Imaging not required for study inclusion).
8. Poorly controlled hypertension
9. Any history of hemorrhagic stroke or lacunar infarct.
10. Current untreated hypothyroidism or thyroid stimulating hormone (TSH)
11. Current history of alcoholism or drug addiction according to the Diagnostic and Statistical Manual of Mental Disorders (DSM) IV criteria within 12 months prior to screening. Use of any illicit drug confirmed by urine toxicology test at screening that would in the opinion of the investigator interfere with study procedures or results.
12. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer resolved by excision, or cervical carcinoma in situ).
13. Any disease or condition that might compromise the hematological, renal, hepatic, pulmonary, endocrine, central nervous, immune, or gastrointestinal systems.
14. Undergoing apheresis or have a planned start of apheresis.
15. Initiation of or change in non-lipid lowering prescription drugs, herbal medicine or supplements (including foods with added plant sterols and stanols) within 6 weeks of screening with the exception of initiation or change in multivitamins used for general health purposes. Short-term use of medications to treat acute conditions, and vaccines are allowed (e.g., antibiotics or allergy medication).
16. History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody (IgG protein) or molecules made of components of monoclonal antibodies (e.g., Enbrel® which contains the Fc portion of an antibody or Lucentis® which is a Fab).
17. Any abnormal hematology values, clinical chemistries, or ECGs at screening judged by the Investigator as clinically significant, which could impact on subject safety, were the potential subject to be included in the study, or interfere with the interpretation of study results.
18. Active phase hepatitis. Stable patients with hepatitis B or C infection >2 years before randomization are eligible.
19. Aspartate transaminase (AST) or alanine transaminase (ALT) > 5 X ULN at screening.
20. Direct bilirubin > 4 X ULN at screening.

22. GFR < 60 mL/min/1.73m2 at screening or undergoing dialysis.

23. Changes in lipid-lowering or antihypertensive medication within 90 days prior to study entry or expected need to modify these medications during study

24. Female subject who has either (1) not used at least 1 highly effective method of birth control for at least 1 month prior to screening or (2) is not willing to use such a method during treatment and for an additional 105 days after the end of treatment, unless the subject is sterilized or postmenopausal.

* Highly effective methods of birth control include not having intercourse or using birth control methods that work at least 99% of the time when used correctly and include: birth control pills, shots, implants or patches, intrauterine devices (IUDs), tubal ligation/occlusion, sexual activity with a male partner who has had a vasectomy, condom or occlusive cap (diaphragm or cervical/vault caps) used with spermicide
* Achieved post-menopausal status is defined as 12 months of spontaneous and continuous amenorrhea in a female

  * 55 years old or 12 months of spontaneous and continuous amenorrhea with a follicle-stimulating hormone (FSH) level > 40 IU/L (or according to the definition of "postmenopausal range" for the laboratory involved in a female <50 years old unless the subject has undergone bilateral oophorectomy.

    25. Pregnant females; breastfeeding females.

    26. Additional exclusion criteria for the FDG-PET/CT imaging (patients with these exclusions may participate in the rest of the trial):

    a. Significant radiation exposure during the year prior to randomization. Significant exposure is defined as i) more than 2 PCI procedures, ii) more than 2 myocardial perfusion studies, or iii) more than 2 CT angiograms.

    b. Any history of radiation therapy.

    c. Current insulin use

    26. Additional exclusion criteria for CTA imaging:
    1. Significant radiation exposure during the year prior to randomization. Significant exposure is defined as i) more than 2 PCI procedures, ii) more than 2 myocardial perfusion studies, or iii) more than 2 CT angiograms (as with FDG-PET/CT).
    2. Any history of radiation therapy (as with FDG-PET/CT).
    3. Any contraindication to beta-blocker (atenolol and metoprolol) or nitroglycerin use, because these drugs are given as part of the standard cardiac CT protocol.
    4. Significant renal dysfunction (defined as an eGFR < 60 mL/min/1.73m2).
    5. Body weight > 300 pounds (136 Kg), because of the CT scanner table limitations.
    6. Allergy to iodine-containing contrast media.
    7. Any history of CABG.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2025-08-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
FDG PET/CT Endpoint | Baseline and Week 52
  Change in Target-to-background ratio from baseline to follow-up study at 52 weeks. The main arterial endpoint is the most diseased segment of the index vessel
FDG PET/CT Endpoint | Baseline Week 24, and 52
  Percent change from baseline in fasting TC, HDL-C, triglycerides, non HDL-C, ApoB, ApoA-I at week 24, and 52
FDG PET/CT Endpoint | Baseline, Week 24, and 52
  Percent change from baseline in fasting oxidized LDL, Lp(a), LpPLA2, sCD14 and T-Cell activation at week 24, and 52
FDG PET/CT Endpoint | Baseline and Week 52
  Correlation of lipid and immune activation parameters to arterial inflammation

SECONDARY OUTCOMES:
Flow mediated vasodilation of the brachial artery (FMD) endpoint | Baseline, Week 24 and Week 52
  Change in FMD from baseline to follow-up at weeks 24, and 52
Flow mediated vasodilation of the brachial artery (FMD) endpoint | Baseline, Week 24 and Week 52
  Correlation of FMD changes to lipid parameters
Flow mediated vasodilation of the brachial artery (FMD) endpoint | Baseline, Week 24 and Week 52
  Correlation of FMD changes to immune parameters
Flow mediated vasodilation of the brachial artery (FMD) endpoint | Baseline Week 24 and Week 52
  Microvascular changes from baseline to weeks 24, and 52
Flow mediated vasodilation of the brachial artery (FMD) endpoint | Baseline, Week 24 and Week 52
  Correlation of microvascular changes to lipid parameters
Flow mediated vasodilation of the brachial artery (FMD) endpoint | Baseline, Week 24 and Week 52
  Correlation of microvascular changes to immune parameters

OTHER OUTCOMES:
Coronary CTA Endpoint | Baseline and Week 52
  Change in non-calcified plaque from baseline to follow-up study at 52 weeks
Coronary CTA Endpoint | Baseline and Week 52
  Change in high-risk plaque from baseline to follow-up study at 52 weeks.
Coronary CTA Endpoint | Baseline and Week 52
  Incidence of new lesions from baseline to follow-up study at 52 weeks
Coronary CTA Endpoint | Baseline and Week 52
  Correlations between change in lipid and change in volume of non-calcified coronary plaque
Coronary CTA Endpoint | Baseline and Week 52
  Correlations between change in lipid and change in high-risk coronary plaque
Coronary CTA Endpoint | Baseline and Week 52
  Correlations between change in immune parameters and change in volume of non-calcified coronary plaque b.change in high-risk coronary plaque
Coronary CTA Endpoint | Baseline and Week 52
  Correlations between change in immune parameters and change in high-risk coronary plaque

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Hsue, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No